CLINICAL TRIAL: NCT05344924
Title: Transarterial Chemoembolization Combined With Penpulimab and Anlotinib for Advanced Hepatocellular Carcinoma：A Nationwide Multicenter Prospective Real-world Study
Brief Title: TACE Combined With Penpulimab and Anlotinib for Advanced HCC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Head of Zhongda Hospital, Zhongda Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHANCE 2205
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Transarterial chemoembolization; Penpulimab; Anlotinib
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Patients in cohort I will receive TACE combined with penpulimab and anlotinib (TACE-A-A Cohort), and patients in cohort II will just receive penpulimab and anlotinib (A-A Cohort).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort I（TACE-A-A Cohort） (Experimental): Patients will receive TACE as needed; penpulimab 200 mg i.v. every 3 weeks(Q3W); and anlotinib 12 mg orally before breakfast,everyday(QD); continue taking for 2 weeks and stop for 1 week, that is, 3 weeks (21 days) as a course of treatment.
  Interventions: Drug: TACE+penpulimab+anlotinib vs. penpulimab+anlotinib
- Cohort II (A-A Cohort) (Experimental): Patients will receive penpulimab 200 mg i.v. every 3 weeks(Q3W); and anlotinib 12 mg orally before breakfast,everyday(QD); continue taking for 2 weeks and stop for 1 week, that is, 3 weeks (21 days) as a course of treatment.
  Interventions: Drug: TACE+penpulimab+anlotinib vs. penpulimab+anlotinib

INTERVENTIONS:
Drug: TACE+penpulimab+anlotinib vs. penpulimab+anlotinib — Patients will receive TACE as needed; penpulimab 200 mg i.v. every 3 weeks(Q3W); and anlotinib 12 mg orally before breakfast,everyday(QD); continue taking for 2 weeks and stop for 1 week, that is, 3 weeks (21 days) as a course of treatment.
  Other Names: The combination of penpulimab+anlotinib with or without TACE

SUMMARY:
The purpose of this multicenter, dual-cohort, prospective real-world study is to explore the efficacy and safety of penpulimab and anlotinib combined with or without TACE, as well as the optimum interval of the combination of penpulimab and anlotinib with TACE in advanced HCC patients.

DETAILED DESCRIPTION:
The efficacy and safety of transarterial chemoembolization (TACE) combined with penpulimab and anlotinib in the treatment of advanced hepatocellular carcinoma (HCC) remain unknown. This is a multicenter, dual-cohort, prospective real-world study with patients receiving normal clinical care. Patients in cohort I will receive TACE combined with penpulimab and anlotinib (TACE-A-A Cohort), and patients in cohort II will just receive penpulimab and anlotinib (A-A Cohort). The primary endpoints of this study are the efficacy of penpulimab and anlotinib combined with or without TACE in advanced HCC patients. While the secondary endpoints include the safety of penpulimab and anlotinib combined with or without TACE, as well as the optimum interval of the combination of penpulimab and anlotinib with TACE in advanced HCC patients. The results will provide further evidence for the clinical practice and the design of future trials.

ELIGIBILITY:
Inclusion criteria:

* Pathologically or clinically diagnosed HCC patients;
* Age of 18-80;
* Barcelona Clinic Liver Cancer (BCLC) stage C (ie, China Liver Cancer Staging (CNLC) stage III);
* with expect survival ≥ 3 months;
* with obtained informed consent;
* will receive penpulimab and anlotinib combined with or without TACE.

Exclusion criteria:

* Contraindications of penpulimab and anlotinib;
* Child-Pugh C;
* Key information (such as imaging, liver function, Eastern Cooperative Oncology Group(ECOG) score, etc.) missing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 2 years
  Time from initiation of either combination therapy to tumor progression according to the modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria or death from any cause.

SECONDARY OUTCOMES:
Objective response rate(ORR) | 2 years
  The proportion of patients with complete response (CR) and partial response (PR) according to the mRECIST criteria.
Overall survival (OS) | up to 5 years
  The time from initiation of either regimen of combination therapy to all-cause death.
Adverse effects | 2 years
  Adverse event (AE)，treatment emergent adverse event(TEAE)，serious adverse event (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital Affiliated to Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No